CLINICAL TRIAL: NCT05898425
Title: Impact of Coronary Collaterals on Intramyocardial Hemorrhage in AMI Patients
Brief Title: Coronary Collaterals and Post-reperfusion Intramyocardial Hemorrhage
Acronym: MIRON-CL
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Rohan Dharmakumar, Executive Director, Krannert Cardiovascular Research Center, Indiana University School of Medicine, Indiana University
Other Study IDs: 19978c
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Coronary Angiography; Intramyocardial Hemorrhage; Cardiac Magnetic Resonance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study examines the relationship between angiographic coronary collaterals (Rentrop grades) and post-reperfusion microvascular injury. This study aims to assess the impact of coronary collateral circulation on intramyocardial hemorrhage incidence and extent.

ELIGIBILITY:
1. Age 18-85 years
2. Index STEMI
3. Coronary angiogram with Primary coronary intervention
4. No contraindications for Cardiac MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises individuals aged 18 years or older who are diagnosed with Index STEMI, based on ACC/AHA criteria, and have completed coronary angiogram with PCI and CMR.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Intramyocardial hemorrhage (IMH) | Day 3
  Collaterals grades (0-III) will be correlated with incidence rate of IMH
Volume of Intramyocardial hemorrhage (IMH) | Day 3
  Collaterals grades (0-III) will be correlated with IMH volume

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Dharmakumar, PhD, Study Director — Indiana University School of Medicine; Keyur P Vora, MD FACC, Principal Investigator — Indiana University School of Medicine
Locations (1):
- IU Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No